CLINICAL TRIAL: NCT03609008
Title: The Effect of Levcromakalim Infusion on the Cranial Arteries Over Several Hours Using a High Resolution MRA Technique in a Randomized, Double-blind Placebo-controlled Design in Healthy Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Levcromakalim & MRI
Record Dates: First submitted 2018-06-26; First posted 2018-08-01 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Dilatation of Cranial Arteries; MMA, STA and MCA; Headache
MeSH Terms: conditions — Headache | interventions — Cromakalim; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind placebo-controlled study with healthy volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Active Comparator): 18 participants will randomly be allocated in a 2:1 order to receive 1 mg levcromakalim or placebo (isotonic saline)
  Interventions: Drug: Levcromakalim
- Saline (Placebo Comparator): 18 participants will randomly be allocated in a 2:1 order to receive 1 mg levcromakalim or placebo (isotonic saline)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — Intravenous administration of levcromakalim or placebo for 20 minutes. To investigate the role of levcromakalim/placebo on cerebral hemodynamic in healthy volunteers.
  Arms: Levcromakalim
Drug: Saline — Intravenous administration of levcromakalim or placebo for 20 minutes. To investigate the role of levcromakalim/placebo on cerebral hemodynamic in healthy volunteers.
  Arms: Saline

SUMMARY:
Healthy participants vill randomly be allocated in a 2:1 order to receive 1 mg levcromakalim or placebo (isotonic saline) for 20 min.

The investigator here examine the effect of levcromakalim infusion on the MMA and the MCA circumference over several hours using a high resolution MRA technique in a randomized, double-blind placebo-controlled design in healthy volunteers. The investigator hypothesized that levcromakalim induces dilatation of cranial arteries.

DETAILED DESCRIPTION:
Healthy participants vill randomly be allocated in a 2:1 order to receive 1 mg levcromakalim or placebo (isotonic saline) for 20 min.

The investigator here examine the effect of levcromakalim infusion on the MMA and the MCA circumference over several hours using a high resolution MRA technique in a randomized, double-blind placebo-controlled design in healthy volunteers. The investigator hypothesized that levcromakalim induces dilatation of cranial arteries.

MR imaging will be performed on a 3.0 Tesla Philips Achieva Scanner (Philips Medical Systems, Best, The Netherlands) using an eight-element phased-array receiver head coil. We will obtain repeated MRA measurements covering the MMA and MCA before and after levcromakalim/placebo infusion

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes.
* 18-60 years.
* 50-100 kg.
* Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

* A history of serious somatic disease
* Migraine or any other type of headache (except episodic tension-type headache less than once a month)
* Daily intake of any medication except contraceptives
* Contraindications for MRI scan.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Change is assessed of cranaial arteries; MMA, STA and MCA | Before and after infusion of levcromakalim compared with before and after infusion of saline. Time of measurements is baseline, 20 min, 110 min, 200 min, 290 min and 350 min after the infusion.
  The investigator will obtain repeated MRA measurements covering the diameter of MMA and MCA before and after levcromakalim/placebo infusion.

SECONDARY OUTCOMES:
Headache | Before (-10 min) and after infusion (+16 hours) of levcromakalim compared with before and after infusion of saline
  Headache intensity will be recorded on a verbal rating scale (VRS) from 0 to 10 (0, no headache; 1, a feeling of pressure; 10, worst imaginable headache).
  Time of headache measurements is before (-10 min) and after infusion (+16 hours) of levcromakalim compared with before and after infusion of saline

CONTACTS AND LOCATIONS:
Locations (1):
- Danish headache center, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Al-Karagholi MA, Ghanizada H, Hansen JM, Skovgaard LT, Olesen J, Larsson HBW, Amin FM, Ashina M. Levcromakalim, an Adenosine Triphosphate-Sensitive Potassium Channel Opener, Dilates Extracerebral but not Cerebral Arteries. Headache. 2019 Oct;59(9):1468-1480. doi: 10.1111/head.13634. Epub 2019 Sep 18. PMID 31535367